CLINICAL TRIAL: NCT01682876
Title: A Phase 3b, Randomized, Observer-Blind, Placebo-Controlled Multi-Center Study Comparing Immunogenicity, Safety and 1 Year Persistence of Antibodies After Either One or Two Doses of Novartis Meningococcal ACWY Conjugate Vaccine, Administered to Healthy Children 2 to 10 Years of Age.
Brief Title: Immunogenicity, Safety and 1 Year Persistence of Antibodies After Either One or Two Doses of Meningococcal ACWY Conjugate Vaccine in Healthy Children 2 Through 10 Years of Age.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 205238; V59_57 (Other: Novartis Vaccines); 2011-004421-27 (EudraCT Number)
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Meningococcal Disease; Infections, Meningococcal
Keywords: Prevention of meningococcal disease, children, vaccine
MeSH Terms: conditions — Meningococcal Infections | interventions — MenACWY-CRM vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 through 5 years (1 Vac) MenACWY-CRM 1 (Placebo Comparator): Subjects 2 through 5 years received one vaccination of MenACWY-CRM
  Interventions: Biological: MenACWY-CRM
- 2 through 5 years (2 Vac) MenACWY-CRM 2 (Active Comparator): Subjects 2 through 5 years received two vaccinations of MenACWY-CRM
  Interventions: Biological: MenACWY-CRM
- 6 through 10 years (1 Vac) MenACWY-CRM 3 (Placebo Comparator): Subjects 6 through 10 years received one vaccination of MenACWY-CRM
  Interventions: Biological: MenACWY-CRM
- 6 through 10 years (2 Vac) MenACWY-CRM 4 (Active Comparator): Subjects 6 through 10 years received two vaccinations of MenACWY-CRM
  Interventions: Biological: MenACWY-CRM

INTERVENTIONS:
Biological: MenACWY-CRM — The investigational meningococcal (groups A, C, Y, and W-135 vaccine) oligosaccharide diphtheria CRM197 conjugate vaccine (MenACWY-CRM) was administered intramuscularly in the nondominant arm

SUMMARY:
This study was designed to conduct a comparative trial to further evaluate the safety, immunogenicity and antibody persistence of two doses of Novartis MenACWY conjugate vaccine, given 2 months apart, versus one dose of Novartis MenACWY conjugate vaccine in children 2 through 10 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children, 2 to 10 years of age who have up to date routine childhood vaccination, according to U.S. ACIP recommendations

Exclusion Criteria:

1. Unwilling or unable to give written informed assent or consent to participate in the study.
2. Perceived to be unreliable or unavailable for the duration of the study period.
3. Previous confirmed or suspected disease caused by N. meningitidis.
4. Previously immunized with a meningococcal vaccine (licensed or investigational).
5. Receipt of any investigational or non-registered product within 30 days prior to enrolment or who expect to receive an investigational drug or vaccine prior to the completion of the study.
6. Receipt or plan to receive any vaccines within 30 days before and after administration of each dose of the study vaccine.

   (certain exceptions influenza vaccines apply)
7. Significant acute infection within the 7 days prior to enrolment or body temperature of 38°C or greater within 3 days prior to enrolment.
8. Previous serious acute, chronic or progressive disease, epilepsy or any progressive neurological disease or history of Guillain-Barre syndrome.
9. History of any anaphylaxis, serious vaccine reactions, or allergy to any vaccine components
10. Impairment/alteration of immune function, either congenital or acquired or resulting from (for example):

    * receipt of immunosuppressive therapy,
    * receipt of immunostimulants,
    * receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives.
11. Known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 715 (Actual)
Dates: Start 2012-10-07 (Actual); Primary Completion 2013-07-02 (Actual); Study Completion 2014-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (18):
- United States (18):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Lake Mary, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Niles, Michigan
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Fremont, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Johnson City, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, West Jordan, Utah

REFERENCES:
- [Derived] Johnston W, Essink B, Kirstein J, Forleo-Neto E, Percell S, Han L, Keshavan P, Smolenov I. Comparative Assessment of a Single Dose and a 2-dose Vaccination Series of a Quadrivalent Meningococcal CRM-conjugate Vaccine (MenACWY-CRM) in Children 2-10 Years of Age. Pediatr Infect Dis J. 2016 Jan;35(1):e19-27. doi: 10.1097/INF.0000000000000931. PMID 26398741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 22 locations
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- 2 Through 5 Years (2 Vac): Subjects 2-5 years of age received two MenACWY-CRM vaccinations
- 2 Through 5 Years (1 Vac): Subjects 2-5 years of age received one MenACWY-CRM vaccination
- 6 Through 10 Years (2 Vac): Subjects 6-10 years of age received two MenACWY-CRM vaccinations
- 6 Through 10 Years (1 Vac): Subjects 6-10 years of age received one MenACWY-CRM vaccination
Period: Overall Study
Arm/Group | 2 Through 5 Years (2 Vac) | 2 Through 5 Years (1 Vac) | 6 Through 10 Years (2 Vac) | 6 Through 10 Years (1 Vac)
Started | 176 | 183 | 180 | 176
Completed | 155 | 163 | 169 | 157
Not Completed | 21 | 20 | 11 | 19
Not completed — Administrative reason | 4 | 4 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 11 | 15 | 9 | 11
Not completed — Protocol Violation | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 2
Not completed — Other | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 Through 5 Years (2 Vac) | 2 Through 5 Years (1 Vac) | 6 Through 10 Years (2 Vac) | 6 Through 10 Years (1 Vac) | Total
Number analyzed (Participants) | 176 | 183 | 180 | 176 | 715
Age, Continuous [Mean (Standard Deviation); unit: year] | 3.5 (1.1) | 3.6 (1.2) | 7.8 (1.4) | 7.8 (1.4) | 5.7 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 88 | 97 | 87 | 356
  Male | 92 | 95 | 83 | 89 | 359

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority of Two Vaccinations Versus One Vaccination of MenACWY-CRM, by Age Cohort, as Measured by the Percentage of Subjects With hSBA Seroresponse Against N. Meningitidis Serogroups A, C, W and Y, at 1 Month After Last Vaccination
Description: Immunogenicity was measured as the percentage of subjects with overall seroresponse and associated 2-sided 97.5% Clopper-Pearson confidence interval (CI), directed against N. meningitidis serogroups A, C, W and Y, by serum bactericidal assay using human complement (hSBA) at 1 month after one vaccination or two vaccinations of MenACWY-CRM given two months apart. Seroresponse is defined as: a. postvaccination hSBA titer ≥1:8 for subjects with a prevaccination hSBA titer <1:4; b. for subjects with a prevaccination hSBA ≥1:4, an increase of at least four times of the prevaccination hSBA titer.
Time Frame: One Month After Last Vaccination ( day 86)
Population: Analysis was done on the primary per-protocol (PP) dataset, i.e. the subjects who received the vaccine correctly; provided evaluable serum samples at the relevant time points; and had no major protocol violations as defined prior to analysis.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | 2 Through 5 Years (2 Vac) | 2 Through 5 Years (1 Vac) | 6 Through 10 Years (2 Vac) | 6 Through 10 Years (1 Vac)
Number analyzed (Participants) | 136 | 144 | 153 | 142
percentage of subjects
  MenA(N=135,143,152,142) | 94 [89 to 97] | 75 [67 to 82] | 89 [83 to 93] | 77 [70 to 84]
  MenC(N=131,140,149,142) | 92 [86 to 96] | 65 [56 to 73] | 93 [87 to 96] | 73 [65 to 80]
  MenW(N=128,135,148,138) | 75 [67 to 82] | 61 [52 to 69] | 58 [50 to 66] | 54 [45 to 62]
  MenY(N=128,133,148,142) | 91 [84 to 95] | 64 [55 to 72] | 89 [83 to 94] | 60 [51 to 68]
Statistical Analysis 1: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); Non-inferiority of seroresponse of two vaccinations vs.one vaccination for age cohort (2 to 5 years of age) for MenA; Test type: Non-Inferiority or Equivalence — Noninferiority was demonstrated for 2 to 5 years of age group if the lower limit of the 2-sided 97.5% confidence interval (CI) for the difference in seroresponse rate between the 2-dose vaccination schedule and the 1-dose vaccination schedule (2-dose schedule minus the 1-dose schedule) was greater than -10% for MenA; MN method; Vaccine Group Differences at Day 86 = 19, 97.5% CI 2-sided [10 to 28.9]
Statistical Analysis 2: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); Non-inferiority of seroresponse of two vaccinations vs. one vaccination for age cohort (2 to 5 years of age) for MenC; Test type: Non-Inferiority or Equivalence — Noninferiority was demonstrated for 2 to 5 years of age group if the lower limit of the 2-sided 97.5% confidence interval (CI) for the difference in seroresponse rate between the 2-dose vaccination schedule and the 1-dose vaccination schedule (2-dose schedule minus the 1-dose schedule) was greater than -10% for MenC; MN method; Vaccine Group Differences at Day 86 = 27, 97.5% CI 2-sided [16.9 to 37.7]
Statistical Analysis 3: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); Non-inferiority of seroresponse of two vaccinations vs. one vaccination for age cohort (2 to 5 years of age) for MenW; Test type: Non-Inferiority or Equivalence — Noninferiority was demonstrated for 2 to 5 years of age group if the lower limit of the 2-sided 97.5% confidence interval (CI) for the difference in seroresponse rate between the 2-dose vaccination schedule and the 1-dose vaccination schedule (2-dose schedule minus the 1-dose schedule) was greater than -10% for MenW; MN method; Vaccine Group Differences at Day 86 = 14, 97.5% CI 2-sided [1.4 to 26.7]
Statistical Analysis 4: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); Non-inferiority of seroresponse of two vaccinations vs. one vaccination for age cohort (2 to 5 years of age) for MenY; Test type: Non-Inferiority or Equivalence — Noninferiority was demonstrated for 2 to 5 years of age group if the lower limit of the 2-sided 97.5% confidence interval (CI) for the difference in seroresponse rate between the 2-dose vaccination schedule and the 1-dose vaccination schedule (2-dose schedule minus the 1-dose schedule) was greater than -10% for Men Y; MN method; Vaccine Group differences at Day 86 = 27, 97.5% CI 2-sided [15.6 to 37.6]
Statistical Analysis 5: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); Non-inferiority of seroresponse of two vaccinations vs. one vaccination for age cohort (6 to 10 years of age) for MenA; Test type: Non-Inferiority or Equivalence — Noninferiority was demonstrated for 6 to 10 years of age group if the lower limit of the 2-sided 97.5% confidence interval (CI) for the difference in seroresponse rate between the 2-dose vaccination schedule and the 1-dose vaccination schedule (2-dose schedule minus the 1-dose schedule) was greater than -10% for MenA; MN method; Vaccines Group Differences at Day 86 = 11, 97.5% CI 2-sided [1.7 to 21.3]
Statistical Analysis 6: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); Non-inferiority of seroresponse of two vaccinations vs. one vaccination for age cohort (6 to 10 years of age) for MenC; Test type: Non-Inferiority or Equivalence — Noninferiority was demonstrated for 6 to 10 years of age group if the lower limit of the 2-sided 97.5% confidence interval (CI) for the difference in seroresponse rate between the 2-dose vaccination schedule and the 1-dose vaccination schedule (2-dose schedule minus the 1-dose schedule) was greater than -10% for MenC; MN method; Vaccines Group differences at Day 86 = 19, 97.5% CI 2-sided [9.9 to 29.2]
Statistical Analysis 7: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); Non-inferiority of seroresponse of two vaccinations vs. one vaccination for age cohort (6 to 10 years of age) for MenW; Test type: Non-Inferiority or Equivalence — Noninferiority was demonstrated for 6 to 10 years of age group if the lower limit of the 2-sided 97.5% confidence interval (CI) for the difference in seroresponse rate between the 2-dose vaccination schedule and the 1-dose vaccination schedule (2-dose schedule minus the 1-dose schedule) was greater than -10% for MenW; MN method; Vaccines Group Differences at Day 86 = 4, 97.5% CI 2-sided [-8.6 to 17.4]
Statistical Analysis 8: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); Non-inferiority of seroresponse for two vaccinations vs. one vaccination for age cohort (6 to 10 years of age) for MenY; Test type: Non-Inferiority or Equivalence — Noninferiority was demonstrated for 6 to 10 years of age group if the lower limit of the 2-sided 97.5% confidence interval (CI) for the difference in seroresponse rate between the 2-dose vaccination schedule and the 1-dose vaccination schedule (2-dose schedule minus the 1-dose schedule) was greater than -10% for MenY; MN method; Vaccines Group Differences at Day 86 = 29, 97.5% CI 2-sided [18.4 to 40]

2. Primary Outcome: Superiority of Two Vaccinations Versus One Vaccination of MenACWY-CRM, by Age Cohort, as Measured by the Percentage of Subjects With hSBA Seroresponse Against N. Meningitidis Serogroups A, C, W and Y, at 1 Month After Last Vaccination
Description: Immunogenicity was measured as the percentage of subjects with overall seroresponse and associated 2-sided 95% CI, directed against N. meningitidis serogroups A, C, W and Y, by hSBA at 1 month after one vaccination or two vaccinations of MenACWY-CRM. Seroresponse -postvaccination hSBA titer ≥1:8 for subjects with a prevaccination hSBA titer <1:4 and for subjects with a prevaccination hSBA ≥1:4, an increase of at least four times of the prevaccination hSBA titer.
Time Frame: One Month After Last Vaccination (day 86)
Population: Analysis was done on the FAS dataset - All subjects in the exposed dataset who provided evaluable serum samples whose assay results were available for at least 1 serogroup on day 1 and 1 post baseline visit.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | 2 Through 5 Years (2 Vac) | 2 Through 5 Years (1 Vac) | 6 Through 10 Years (2 Vac) | 6 Through 10 Years (1 Vac)
Number analyzed (Participants) | 159 | 165 | 172 | 163
percentage of subjects
  MenA(N=158,163,171,163) | 95 [90 to 98] | 77 [69 to 83] | 89 [84 to 94] | 79 [71 to 85]
  MenC(N=154,157,167,162) | 93 [88 to 96] | 65 [57 to 72] | 93 [89 to 97] | 75 [68 to 82]
  MenW(N=150,154,167,159) | 75 [68 to 82] | 61 [53 to 69] | 57 [49 to 65] | 52 [44 to 60]
  MenY(N=150,153,167,163) | 90 [84 to 94] | 62 [54 to 70] | 89 [83 to 93] | 60 [52 to 68]
Statistical Analysis 1: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); Superiority for age cohort (2 through 5 years of age) for MenA was demonstrated if the lower limit of the 2-sided (1-2α) % CI for seroresponse increase between the 2-dose vaccination schedule and the 1-dose vaccination schedule was above 10% for MenA; Test type: Superiority or Other; MN method; Vaccine Group Differences at Day 86 = 18, 98.75% CI 2-sided [9.1 to 28]
Statistical Analysis 2: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); Superiority for age cohort (2 through 5 years of age) for MenC was demonstrated if the lower limit of the 2-sided (1-2α) % CI for seroresponse increase between the 2-dose vaccination schedule and the 1-dose vaccination schedule was above 10% for MenC; Test type: Superiority or Other; MN method; Vaccine Group Differences at Day 86 = 28, 98.75% CI [17.1 to 38.7]
Statistical Analysis 3: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); Superiority for age cohort (2 through 5 years of age) for MenW was demonstrated if the lower limit of the 2-sided (1-2α) % CI for seroresponse increase between the 2-dose vaccination schedule and the 1-dose vaccination schedule was above 10% for MenW; Test type: Superiority or Other; MN method; Vaccine Group differences at Day 86 = 14, 98.75% CI 2-sided [1 to 27.1]
Statistical Analysis 4: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); Superiority for age cohort (2 through 5 years of age) for MenY was demonstrated if the lower limit of the 2-sided (1-2α) % CI for seroresponse increase between the 2-dose vaccination schedule and the 1-dose vaccination schedule was above 10% for MenY; Test type: Superiority or Other; MN method; Vaccine groups Differences at Day 86 = 28, 98.75% CI 2-sided [16.2 to 39.3]
Statistical Analysis 5: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); Superiority for age cohort (6 through 10 years of age) for MenA was demonstrated if the lower limit of the 2-sided (1-2α) % CI for seroresponse increase between the 2-dose vaccination schedule and the 1-dose vaccination schedule was above 10% for MenA; Test type: Superiority or Other; MN method; Vaccine groups differences at Day 86 = 11, 98.75% CI 2-sided [1 to 21.2]
Statistical Analysis 6: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); Superiority for age cohort (6 through 10 years of age) for MenC was demonstrated if the lower limit of the 2-sided (1-2α) % CI for seroresponse increase between the 2-dose vaccination schedule and the 1-dose vaccination schedule was above 10% for MenC; Test type: Superiority or Other; MN method; Vaccine Group differences at Day 86 = 18, 97.5% CI 2-sided [9.5 to 27.1]
Statistical Analysis 7: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); Superiority for age cohort (6 through 10 years of age) for MenW was demonstrated if the lower limit of the 2-sided (1-2α) % CI for seroresponse increase between the 2-dose vaccination schedule and the 1-dose vaccination schedule was above 10% for MenW; Test type: Superiority or Other; MN method; Vaccine Group Differences at Day 86 = 5, 98.75% CI 2-sided [-8.4 to 18.8]
Statistical Analysis 8: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); Superiority for age cohort (6 through 10 years of age) for MenY was demonstrated if the lower limit of the 2-sided (1-2α) % CI for seroresponse increase between the 2-dose vaccination schedule and the 1-dose vaccination schedule was above 10% for MenY; Test type: Superiority or Other; MN method; Vaccine group Differences at Day 86 = 29, 98.75% CI 2-sided [17 to 39.6]

3. Secondary Outcome: Percentage of Subjects With hSBA Titer ≥1:8, Directed Against N. Meningitidis Serogroups A, C, W and Y At One Month After One or Two Vaccination(s) of MenACWY-CRM
Description: Immunogenicity was measured as the percentage of subjects who achieved hSBA titer ≥1:8 and associated 95% CI, at one month after one vaccination or two vaccinations of MenACWY-CRM.
Time Frame: One Month After Last Vaccination (day 86)
Population: Analysis was done on the primary PP dataset.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | 2 Through 5 Years (2 Vac) | 2 Through 5 Years (1 Vac) | 6 Through 10 Years (2 Vac) | 6 Through 10 Years (1 Vac)
Number analyzed (Participants) | 136 | 144 | 153 | 142
percentage of subjects
  MenA(N=135,143,152,142) | 95 [90 to 98] | 76 [68 to 82] | 91 [85 to 95] | 80 [73 to 86]
  MenC(N=131,140,149,142) | 98 [95 to 100] | 76 [68 to 83] | 99 [95 to 100] | 89 [82 to 93]
  MenW(N=128,135,148,138) | 99 [96 to 100] | 92 [86 to 96] | 99 [96 to 100] | 96 [91 to 98]
  MenY(N=128,133,148,142) | 96 [91 to 99] | 69 [61 to 77] | 96 [91 to 98] | 73 [64 to 80]

4. Secondary Outcome: Geometric Mean Titers of Subjects, Directed Against N. Meningitidis Serogroups A, C, W and Y At One Month After One or Two Vaccination(s) of MenACWY-CRM
Description: Immunogenicity was measured as hSBA geometric mean titers (GMTs) and 95% CI against N. meningitidis serogroups A, C, W and Y, one month after one vaccination or two vaccinations of MenACWY-CRM.
Time Frame: One Month After Last Vaccination (day 86)
Population: Analysis was done on the primary PP dataset
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 2 Through 5 Years (2 Vac) | 2 Through 5 Years (1 Vac) | 6 Through 10 Years (2 Vac) | 6 Through 10 Years (1 Vac)
Number analyzed (Participants) | 136 | 144 | 153 | 142
Titer
  MenA(N=135,143,152,142) | 68 [54 to 86] | 21 [17 to 27] | 67 [52 to 87] | 36 [28 to 47]
  MenC(N=131,140,149,142) | 146 [115 to 186] | 22 [18 to 28] | 165 [126 to 217] | 67 [51 to 89]
  MenW(N=128,135,148,138) | 191 [150 to 243] | 104 [83 to 132] | 169 [138 to 206] | 95 [78 to 117]
  MenY(N=128,133,148,142) | 70 [55 to 90] | 15 [12 to 19] | 76 [58 to 99] | 26 [20 to 34]

5. Secondary Outcome: Percentage of Subjects With hSBA Titer ≥1:8, Directed Against N. Meningitidis Serogroups A, C, W and Y At One Year After One or Two Vaccination(s) of MenACWY-CRM
Description: Immunogenicity was measured as the percentage of subjects with hSBA titer ≥1:8 and associated 95% CI at one year after one vaccination or two vaccinations of MenACWY-CRM.
Time Frame: One year after one vaccination or two vaccinations (day 422).
Population: Analysis was done on the persistence PP dataset
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | 2 Through 5 Years (2 Vac) | 2 Through 5 Years (1 Vac) | 6 Through 10 Years (2 Vac) | 6 Through 10 Years (1 Vac)
Number analyzed (Participants) | 136 | 144 | 153 | 142
percentages of subjects
  MenA(N=122,131,142,130) | 30 [22 to 39] | 11 [6 to 17] | 30 [22 to 38] | 20 [14 to 28]
  MenC(N=123,128,141,130) | 61 [52 to 70] | 41 [32 to 50] | 81 [73 to 87] | 55 [46 to 64]
  MenW(N=121,127,139,130) | 92 [85 to 96] | 91 [84 to 95] | 94 [89 to 97] | 90 [84 to 95]
  MenY(N=121,122,140,130) | 67 [58 to 75] | 57 [48 to 66] | 75 [67 to 82] | 65 [57 to 74]

6. Secondary Outcome: Geometric Mean Titers of Subjects, Directed Against N. Meningitidis Serogroups A, C, W and Y At One Year After One or Two Vaccination(s) of MenACWY-CRM
Description: Immunogenicity was measured as hSBA GMTs and 95% CI against N. meningitidis serogroups A, C, W and Y at one year after one vaccination or two vaccinations of MenACWY-CRM.
Time Frame: One year after one vaccination or two vaccinations (day 422).
Population: Analysis was done on the persistence PP dataset
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 2 Through 5 Years (2 Vac) | 2 Through 5 Years (1 Vac) | 6 Through 10 Years (2 Vac) | 6 Through 10 Years (1 Vac)
Number analyzed (Participants) | 136 | 144 | 153 | 142
Titers
  MenA(N=122,131,142,130) | 4.72 [3.91 to 5.71] | 2.66 [2.22 to 3.19] | 4.66 [3.75 to 5.81] | 3.56 [2.84 to 4.46]
  MenC(N=123,128,141,130) | 10 [8.34 to 13] | 7.03 [5.63 to 8.76] | 24 [18 to 31] | 15 [12 to 20]
  MenW(N=121,127,139,130) | 49 [39 to 62] | 39 [31 to 49] | 64 [52 to 79] | 47 [38 to 59]
  MenY(N=121,122,140,130) | 14 [11 to 17] | 9.88 [7.8 to 13] | 20 [15 to 25] | 13 [9.96 to 16]

7. Secondary Outcome: Number of 2 to 5 Years-Old Subjects Who Reported Solicited Local and Systemic Adverse Events After Any Vaccination
Description: Safety was assessed as the number of 2 to 5 years-old subjects who reported solicited local and systemic adverse events from day 1 up to and including day 7 after one or two vaccination(s) of MenACWY-CRM
Time Frame: From Days 1-7 after each vaccination
Population: Analysis was done on the safety dataset i.e. the subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: subjects
Arm/Group | 2 Through 5 Years (2 Vac) | 2 Through 5 Years (1 Vac)
Number analyzed (Participants) | 176 | 182
subjects
  Erythema(N=173,175) | 25 | 11
  Induration(N=173,175) | 19 | 7
  Tenderness (N=174,175) | 84 | 79
  Change in Eating Habits(N=173,175) | 26 | 30
  Sleepiness(N=173,175) | 49 | 46
  Irritability(N=173,175) | 51 | 50
  Body Temperature >=38.0(N=174,175) | 9 | 12
Statistical Analysis 1: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced erythema in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 2.3, 95% CI 2-sided [1.17 to 4.53]
Statistical Analysis 2: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced induration in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 2.75, 95% CI 2-sided [1.18 to 6.36]
Statistical Analysis 3: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced tenderness in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.85 to 1.34]
Statistical Analysis 4: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced change in eating habits in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.54 to 1.42]
Statistical Analysis 5: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced sleepiness in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.76 to 1.52]
Statistical Analysis 6: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced irritability in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.74 to 1.43]
Statistical Analysis 7: Comparison: 2 Through 5 Years (2 Vac) vs 2 Through 5 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced fever (≥38 °C) in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.33 to 1.74]

8. Secondary Outcome: Numbers of 6 to 10 Years-Old Subjects Who Reported Solicited Local and Systemic Adverse Events After Any Vaccination
Description: Safety was assessed as the number of 6 to 10 years-old subjects who reported solicited local and systemic adverse events from day 1 up to and including day 7 after one or two vaccination(s) of MenACWY-CRM
Time Frame: From Days 1-7 after each vaccination
Population: Analysis was done on the safety dataset
Measure: Number; unit: Subjects
Arm/Group | 6 Through 10 Years (2 Vac) | 6 Through 10 Years (1 Vac)
Number analyzed (Participants) | 180 | 175
Subjects
  Erythema(N=178,166) | 23 | 15
  Induration(N=178,166) | 24 | 15
  Pain(N=178,166) | 106 | 78
  Loss of Appetite(N=177,166) | 27 | 14
  Nausea(N=177,165) | 29 | 21
  Fatigue(N=177,166) | 44 | 25
  Myalgia(N=177,165) | 63 | 43
  Arthralgia(N=177,165) | 20 | 9
  Headache(N=177,165) | 55 | 28
  Body Temperature>=38.0(N=178,166) | 11 | 9
Statistical Analysis 1: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; Risk Ratio (RR) = 1.43, 95% CI 2-sided [0.77 to 2.65]
Statistical Analysis 2: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; Risk Ratio (RR) = 1.49, 95% CI 2-sided [0.81 to 2.74]
Statistical Analysis 3: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced pain in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 1.27, 95% CI 2-sided [1.04 to 1.55]
Statistical Analysis 4: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced loss of appetite in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 1.81, 95% CI 2-sided [0.98 to 3.33]
Statistical Analysis 5: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced nausea in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 1.29, 95% CI 2-sided [0.77 to 2.17]
Statistical Analysis 6: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced fatigue in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 1.65, 95% CI 2-sided [1.06 to 2.57]
Statistical Analysis 7: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced myalgia in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 1.37, 95% CI 2-sided [0.99 to 1.89]
Statistical Analysis 8: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced arthralgia in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 2.07, 95% CI 2-sided [0.97 to 4.42]
Statistical Analysis 9: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); The safety of two vaccine groups was compared by calculating risk ratio of the proportions of subjects who experienced headache in the two doses versus in the one dose of MenACWY-CRM; Test type: Superiority or Other; Risk Ratio (RR) = 1.83, 95% CI 2-sided [1.22 to 2.74]
Statistical Analysis 10: Comparison: 6 Through 10 Years (2 Vac) vs 6 Through 10 Years (1 Vac); [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.48 to 2.68]

9. Secondary Outcome: Number of Subjects Who Reported Selected AEs After Any Vaccination
Description: Safety was assessed as the number subjects who reported Selected AEs from day 1 up to day 86 after one or two vaccination(s) of MenACWY-CRM
Time Frame: Day 1 to Day 86
Population: Analysis was done on Safety Set Unsolicited AEs
Measure: Number; unit: Subjects
Arm/Group | 2 Through 5 Years (2 Vac) | 2 Through 5 Years (1 Vac) | 6 Through 10 Years (2 Vac) | 6 Through 10 Years (1 Vac)
Number analyzed (Participants) | 179 | 179 | 181 | 174
Subjects
  SAEs | 1 | 0 | 0 | 0
  At least possibly related SAEs | 0 | 0 | 0 | 0
  Medically attended AEs | 50 | 55 | 46 | 46
  At least possibly related medically attended AEs | 0 | 3 | 1 | 1
  AEs resulting in premature withdrawal | 0 | 0 | 0 | 1
  Deaths | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Subjects Who Reported Selected AEs After Any Vaccination
Description: Safety was assessed as the number subjects who reported Selected AEs from day 1 up to day 422 after one or two vaccination(s) of MenACWY-CRM
Time Frame: Day 1 to Day 422
Population: Analysis was done on safety set
Measure: Number; unit: Subjects
Arm/Group | 2 Through 5 Years (2 Vac) | 2 Through 5 Years (1 Vac) | 6 Through 10 Years (2 Vac) | 6 Through 10 Years (1 Vac)
Number analyzed (Participants) | 179 | 179 | 181 | 174
Subjects
  Medically attended AEs | 103 | 101 | 95 | 97
  At least possibly related medically attended AEs | 1 | 4 | 1 | 2
  AEs resulting in premature withdrawal | 0 | 0 | 0 | 1
  SAEs | 2 | 1 | 1 | 1
  Deaths | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout study period
Description: Serious adverse events (SAEs) were collected from day 1 to study termination/early termination.
Groups:
- Total: Total Population
Arm/Group | 2 Through 5 Years (2 Vac) | 2 Through 5 Years (1 Vac) | 6 Through 10 Years (2 Vac) | 6 Through 10 Years (1 Vac) | Total
Serious Adverse Events (participants affected / at risk) | 2/179 | 1/179 | 1/181 | 1/174 | 5/713
Other Adverse Events (participants affected / at risk) | 148/179 | 142/179 | 153/181 | 133/174 | 576/713
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 Through 5 Years (2 Vac) (N=179) | 2 Through 5 Years (1 Vac) (N=179) | 6 Through 10 Years (2 Vac) (N=181) | 6 Through 10 Years (1 Vac) (N=174) | Total (N=713)
IMMUNE THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
OTITIS MEDIA (Infections and infestations) | 1 | 0 | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
PETIT MAL EPILEPSY (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
INTERMITTENT EXPLOSIVE DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
OPPOSITIONAL DEFIANT DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2 Through 5 Years (2 Vac) (N=179) | 2 Through 5 Years (1 Vac) (N=179) | 6 Through 10 Years (2 Vac) (N=181) | 6 Through 10 Years (1 Vac) (N=174) | Total (N=713)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 | 6 | 5 | 9 | 24
DIARRHOEA (Gastrointestinal disorders) | 8 | 10 | 5 | 5 | 28
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 29 | 23 | 52
VOMITING (Gastrointestinal disorders) | 19 | 19 | 15 | 11 | 64
FATIGUE (General disorders) | 1 | 1 | 47 | 32 | 81
INJECTION SITE ERYTHEMA (General disorders) | 71 | 48 | 64 | 49 | 232
INJECTION SITE INDURATION (General disorders) | 54 | 39 | 60 | 40 | 193
INJECTION SITE PAIN (General disorders) | 93 | 91 | 120 | 88 | 392
PYREXIA (General disorders) | 29 | 34 | 26 | 26 | 115
CONJUNCTIVITIS (Infections and infestations) | 7 | 11 | 1 | 3 | 22
EAR INFECTION (Infections and infestations) | 15 | 6 | 5 | 3 | 29
NASOPHARYNGITIS (Infections and infestations) | 2 | 11 | 4 | 4 | 21
OTITIS MEDIA (Infections and infestations) | 19 | 24 | 7 | 8 | 58
PHARYNGITIS (Infections and infestations) | 16 | 16 | 18 | 6 | 56
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 12 | 18 | 17 | 14 | 61
SINUSITIS (Infections and infestations) | 8 | 12 | 6 | 8 | 34
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 22 | 21 | 13 | 16 | 72
VIRAL INFECTION (Infections and infestations) | 9 | 13 | 7 | 4 | 33
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 1 | 27 | 16 | 45
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 22 | 13 | 35
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 66 | 48 | 114
HEADACHE (Nervous system disorders) | 6 | 8 | 62 | 38 | 114
SOMNOLENCE (Nervous system disorders) | 54 | 48 | 0 | 1 | 103
EATING DISORDER (Psychiatric disorders) | 26 | 30 | 0 | 0 | 56
IRRITABILITY (Psychiatric disorders) | 55 | 51 | 1 | 1 | 108
COUGH (Respiratory, thoracic and mediastinal disorders) | 22 | 17 | 12 | 15 | 66
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 2 | 10 | 3 | 1 | 16
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 14 | 9 | 3 | 5 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less